CLINICAL TRIAL: NCT03814889
Title: Passive Tactile Stimulation for Stroke Rehabilitation
Acronym: PTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Allison Okamura, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49330
Record Dates: First submitted 2019-01-16; First posted 2019-01-24 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Stroke; Stroke, Ischemic; Stroke Hemorrhagic; Spasticity as Sequela of Stroke
Keywords: spasticity; tone; hemiplegia; hemiparesis; arm; hand; vibration
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Muscle Spasticity; Hemiplegia; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Acute Stimulation: Vibration pattern 1-3 and sham control (Active Comparator): All participants try on several wearable prototypes in our laboratory that provide vibration or sham stimulation to the arm. Sensors or electrodes taped onto the arm and hand will sense muscle activity and record any changes during periods of vibration and periods with vibration turned off.
  Interventions: Device: Vibration pattern; Device: No vibration
- Longitudinal Stimulation: Vibration pattern 4 (Active Comparator): 1) If the patient gets Botox injections in their hand and arm, their arm function will be measured for three months during this standard care. 2) Next, all patients will be given a wearable device to take home. The patient will wear the device while feeling vibrations for 3 hours during the day while awake for two months. During this time and 1 month after this intervention, arm function will be tested.
  Interventions: Device: Vibration pattern

INTERVENTIONS:
Device: Vibration pattern — Vibration patterns applied to the affected limb based on pilot study results.
Device: No vibration — These patients will wear a glove with a blinking light instead of feeling vibrations.
  Arms: Acute Stimulation: Vibration pattern 1-3 and sham control

SUMMARY:
Stroke can lead to weakness and spasticity in the arm or hand. The purpose of this study is to optimize the design of gentle vibratory stimulation delivered to the hands of individuals with chronic stroke, and explore the effect on range of movement and spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older.
* diagnosis of stroke with upper extremity spasticity or other movement deficits that affect strength and range of movement.
* willing to participate in the vibrotactile stimulation sessions for consecutive days and willing to return for follow up visits as needed for the PHASE in progress.
* able to provide informed consent.

Exclusion Criteria:

* Patients with severe contracture that precludes Modified Ashworth Score (MAS) testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison M Okamura, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Neuroscience Health Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Seim C, Chen B, Han C, Vacek D, Wu LS, Lansberg M, Okamura A. Relief of post-stroke spasticity with acute vibrotactile stimulation: controlled crossover study of muscle and skin stimulus methods. Front Hum Neurosci. 2023 Aug 29;17:1206027. doi: 10.3389/fnhum.2023.1206027. eCollection 2023. PMID 37706171

RESULTS

PARTICIPANT FLOW:
Groups:
- Acute Stimulation: Vibration Pattern 1-3 and Sham Control: All participants try on several wearable prototypes in our laboratory that provide vibration to the arm. Sensors or electrodes taped onto the arm and hand will sense muscle activity and record any changes during periods of vibration and periods with vibration turned off.
Period: Acute Testing
Arm/Group | Acute Stimulation: Vibration Pattern 1-3 and Sham Control | Longitudinal Stimulation: Vibration Pattern 4
Started | 14 | 0
Completed | 14 | 0
Not Completed | 0 | 0
Period: Longitudinal Testing
Arm/Group | Acute Stimulation: Vibration Pattern 1-3 and Sham Control | Longitudinal Stimulation: Vibration Pattern 4
Started | 0 | 21
Completed | 0 | 20
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Acute Stimulation: Vibration Patterns 1-3 and Sham Control: All participants try on several wearable prototypes in our laboratory that provide vibration to the arm. Sensors or electrodes taped onto the arm and hand will sense muscle activity and record any changes during periods of vibration and periods with vibration turned off.
- Total: Total of all reporting groups
Arm/Group | Acute Stimulation: Vibration Patterns 1-3 and Sham Control | Longitudinal Stimulation: Vibration Pattern 4 | Total
Number analyzed (Participants) | 14 | 21 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (10.3) | 54.4 (13.2) | 56.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 14 | 19
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 14 | 20 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 12 | 18
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 21 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Ashworth at 12 Weeks
Description: Modified Ashworth Scale (from https://www.sralab.org/rehabilitation-measures/ashworth-scale-modified-ashworth-scale). Lower Modified Ashworth scale values indicate a better outcome.
  Measures spastic hypertonia by manually moving an affected joint at set velocities.
  Scores:
  0 (0) - No increase in muscle tone
  1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM (range of movement) 2 (3) - More marked increase in musce tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Time Frame: Change from Baseline Modified Ashworth at 12 weeks
Population: This measure was conducted on only one group.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Acute Stimulation: Vibration Patterns 1-3 and Sham Control | Longitudinal Stimulation: Vibration Pattern 4
Number analyzed (Participants) | 0 | 20
units on a scale |  | 1.1 (0.22)
Statistical Analysis 1: Comparison: Longitudinal Stimulation: Vibration Pattern 4; Test type: Other; p = 0.00025, Wilcoxon Signed-Rank; Paired, ordinal data

2. Primary Outcome: Change in Modified Ashworth at 8 Weeks
Description: Modified Ashworth Scale (from https://www.sralab.org/rehabilitation-measures/ashworth-scale-modified-ashworth-scale) Lower Modified Ashworth scale values indicate a better outcome.
  Measures spastic hypertonia by manually moving an affected joint at set velocities.
  Scores:
  0 (0) - No increase in muscle tone
  1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM (range of movement) 2 (3) - More marked increase in musce tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Time Frame: Change from Baseline Modified Ashworth at 8 weeks
Population: This measure was conducted on only one group.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Vibration Patterns 1-3 and Sham Control: All participants try on several wearable prototypes in our laboratory that provide vibration to the arm. Sensors or electrodes taped onto the arm and hand will sense muscle activity and record any changes during periods of vibration and periods with vibration turned off.
- Vibration Pattern 4: 1) If the patient gets Botox injections in their hand and arm, their arm function will be measured for three months during this standard care. 2) Next, all patients will be given a wearable device to take home. The patient will wear the device while feeling vibrations for 3 hours during the day while awake for two months. During this time and 1 month after this intervention, arm function will be tested.
Arm/Group | Vibration Patterns 1-3 and Sham Control | Vibration Pattern 4
Number analyzed (Participants) | 0 | 20
units on a scale |  | 0.9 (0.28)
Statistical Analysis 1: Comparison: Vibration Pattern 4; Test type: Other; p = 0.0014, Wilcoxon Signed-Rank

3. Primary Outcome: Change in Range of Motion at 8 Weeks
Description: Finger extension range.
Time Frame: Change from Baseline Range of Motion at 8 weeks
Population: This measure was conducted on only one group.
Measure: Mean (Standard Error); unit: degrees of finger extension
Groups:
- Vibration Patterns 1-3 and Sham Control; Vibration Pattern 4: All participants try on several wearable prototypes in our laboratory that provide vibration to the arm. Sensors or electrodes taped onto the arm and hand will sense muscle activity and record any changes during periods of vibration and periods with vibration turned off.
  1) If the patient gets Botox injections in their hand and arm, their arm function will be measured for three months during this standard care. 2) Next, all patients will be given a wearable device to take home. The patient will wear the device while feeling vibrations for 3 hours during the day while awake for two months. During this time and 1 month after this intervention, arm function will be tested.
Arm/Group | Vibration Patterns 1-3 and Sham Control | Vibration Pattern 4
Number analyzed (Participants) | 0 | 20
degrees of finger extension |  | 11.6 (5.2)
Statistical Analysis 1: Comparison: Vibration Pattern 4; Test type: Other; p = 0.02, t-test, 1 sided

4. Primary Outcome: Change in Range of Motion at 12 Weeks
Description: Finger extension range.
Time Frame: Change from Baseline Range of Motion at 12 weeks
Population: This measure was conducted on only one group.
Measure: Mean (Standard Error); unit: degrees of finger extension
Arm/Group | Vibration Patterns 1-3 and Sham Control | Vibration Pattern 4
Number analyzed (Participants) | 0 | 20
degrees of finger extension |  | 18.4 (4.3)
Statistical Analysis 1: Comparison: Vibration Pattern 4; Test type: Other; p = 0.001, t-test, 1 sided

5. Primary Outcome: Change in Modified Ashworth During Stimulation (Pattern 1).
Description: as for outcome 1
Time Frame: 20 minutes after stimulation start
Population: This measure was only taken for one group of patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Vibration Pattern 1-3 and Sham Control: All participants try on several wearable prototypes in our laboratory that provide vibration to the arm. Sensors or electrodes taped onto the arm and hand will sense muscle activity and record any changes during periods of vibration and periods with vibration turned off.
Arm/Group | Vibration Pattern 1-3 and Sham Control | Vibration Pattern 4
Number analyzed (Participants) | 14 | 0
units on a scale | 0.39 (0.96) |

6. Primary Outcome: Change in Modified Ashworth During Stimulation (Pattern 2).
Description: as for outcome 1
Time Frame: 20 minutes after stimulation start
Population: This measure was only taken for one group of patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vibration Pattern 1-3 and Sham Control | Vibration Pattern 4
Number analyzed (Participants) | 14 | 0
units on a scale | 0.25 (0.86) |

7. Primary Outcome: Change in Modified Ashworth During Stimulation (Pattern 3).
Description: as for outcome 1
Time Frame: 20 minutes after stimulation start
Population: This measure was only taken for one group of patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vibration Pattern 1-3 and Sham Control | Vibration Pattern 4
Number analyzed (Participants) | 14 | 0
units on a scale | 1.11 (0.84) |
Statistical Analysis 1: Comparison: Vibration Pattern 1-3 and Sham Control; Test type: Other; p = 0.001, Wilcoxcon Signed-Ranks

8. Primary Outcome: Change in Modified Ashworth During Stimulation (Sham Control).
Description: as for outcome 1
Time Frame: 20 minutes after stimulation start
Population: This measure was only taken for one group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vibration Pattern 1-3 and Sham Control | Vibration Pattern 4
Number analyzed (Participants) | 14 | 0
units on a scale | 0 (0.56) |

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed up to one month for Vibration Pattern 1-3 and Sham Control Arms and up to three-six months for Vibration Pattern 4 Arm
Groups:
- Vibration Pattern 1; Vibration Pattern 2; Vibration Pattern 3; Sham Control: All participants try on several wearable prototypes in our laboratory that provide vibration to the arm. Sensors or electrodes taped onto the arm and hand will sense muscle activity and record any changes during periods of vibration and periods with vibration turned off.
Arm/Group | Vibration Pattern 1 | Vibration Pattern 2 | Vibration Pattern 3 | Sham Control | Vibration Pattern 4
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/21
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT03814889/Prot_SAP_000.pdf